CLINICAL TRIAL: NCT04873531
Title: Feasibility of Neostigmine as a Reversal Agent of Neuromuscular Blockade for Intraoperative Neuromonitoring During Thyroid Surgery: a Prospective Randomized Controlled Study
Brief Title: Feasibility of Neostigmine for Intraoperative Neuromonitoring in Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-2021-12
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Thyroid Diseases; Surgical Injury; Nerve Monitoring
Keywords: thyroid surgery; recurrent laryngeal nerve; neostigmine; intraoperative neuromonitoring
MeSH Terms: conditions — Thyroid Diseases; Intraoperative Complications | interventions — Neostigmine; Saline Solution

STUDY DESIGN:
Intervention Model Description: a randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: For participant, they will be blind to the group which they will be assigned. The surgeon, who will evaluate the quality of the signal, will be blinded to patient's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neostigmine (Experimental): For the Neostigmine (N) group, neostigmine (0.03 mcg / kg) and glycopyrrolate with a 5:1 ratio will be administered just after tracheal intubation.
  Investigators evaluate the quality of signal of IONM during the surgery.
  Interventions: Drug: Neostigmine
- Normal saline (Placebo Comparator): For the Normal saline (NS) group, normal saline with a same volume of the N group will be administered just after tracheal intubation.
  Investigators evaluate the quality of signal of IONM during the surgery.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Neostigmine — For the N group, neostigmine (0.03 mcg / kg) and glycopyrrolate with a 5:1 ratio will be administered just after tracheal intubation.
  Investigators evaluate the quality of signal of IONM during the surgery.
  Other Names: N group
  Arms: Neostigmine
Drug: Normal saline — For the NS group, neostigmine normal saline (0.09 cc/kg; the same volume of the group N) will be administered just after tracheal intubation.
  Investigators evaluate the quality of signal of IONM during the surgery.
  Other Names: NS group
  Arms: Normal saline

SUMMARY:
For successful intraoperative neuromonitoring (IONM), adequate reversal of neuromuscular blocking agent is a prerequisite in thyroid surgery with .

The aim of this study is to investigate the feasibility of neostigmine just after tracheal intubation on the IONM in thyroid surgery.

DETAILED DESCRIPTION:
For successful intraoperative neuromonitoring (IONM), adequate reversal of neuromuscular blocking agent is a prerequisite in thyroid surgery with .

The aim of this study is to investigate the feasibility of neostigmine just after tracheal intubation on the IONM in thyroid surgery.

This study will be performed as a randomized controlled trial with two groups (N group: neostigmine group and NS group: normal saline group).

For the N group, neostigmine (0.03 mcg / kg) and glycopyrrolate with a 5:1 ratio will be administered just after tracheal intubation.

For the NS group, normal saline with a same volume of the N group will be administered just after tracheal intubation.

For all patients of two groups, investigators evaluate the quality of signal of IONM during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* open thyroid surgery with intraoperative neuromonitoring

Exclusion Criteria:

* refusal to participate in the study
* rocuronium should not be used (e.g. renal dysfunction patient)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Time to recovery of cricothyroid muscle twitching | perioperative
  Time from the rocuronium administration to recovery of cricothyroid muscle twitching

SECONDARY OUTCOMES:
amplitude of EMG for V1 | During surgery
  micro-volts (uV), Electromyography amplitude of the vagus nerve before tumor manipulation
amplitude of EMG for R1 | During surgery
  micro-volts (uV), Electromyography amplitude of the recurrent laryngeal nerve before tumor manipulation
amplitude of EMG for R2 | During surgery
  micro-volts (uV), Electromyography amplitude of the recurrent laryngeal nerve after tumor removal
amplitude of EMG for V2 | During surgery
  micro-volts (uV), Electromyography amplitude of the vagus nerve after tumor removal
number of patients with involuntary movements disrupting surgery | During surgery
  number, number of patients who move involuntarily during surgery, which disrupt and pause the surgery to prevent harmful events, such as tracheal injuries by a sharp surgical devices during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, MD.PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
possible, If there would be reasonable explanation for sharing